CLINICAL TRIAL: NCT06285110
Title: HIV-1 Subtype-specific Drug Resistance in Patients Failing Dolutegravir-based 1st, 2nd or 3rd Line Regimens: the International Epidemiological Databases to Evaluate AIDS (IeDEA)
Brief Title: HIV-1 Subtype-specific Drug Resistance in Patients Failing Dolutegravir (DTG) Based Regimen
Acronym: DTG-Resist
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: University of Zurich (Other); ETH Zurich (Other); University of KwaZulu (Other); University of Bristol (Other)
Responsible Party: Sponsor
Other Study IDs: DTG Resist
Record Dates: First submitted 2023-05-08; First posted 2024-02-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hiv
Keywords: HIV; Dolutegravir drug resistance mutations; Virologic failure; DTG based regimen
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People living with HIV: People living with HIV and on a Dolutegravir-based ART regimen, and experiencing treatment failure.

SUMMARY:
This is a prospective observational study enrolling People Living with HIV (PLHIV) who are on a Dolutegravir-based AntiRetroviral Treatment (ART) regimen and experiencing virologic failure. Virologic failure is defined as two consecutive viral load measurements of >1000 copies/mL of blood. The main aim of the study is to identify the drug-resistance mutations in the viral genome that are associated with this failure.

To achieve this goal, patients fulfilling the eligibility criteria will be invited for a single study visit for the collection of blood. The extracted HIV virus will be sequenced through whole genome sequencing methods to identify the drug-resistance mutations. The study is conducted in 15-20 countries within six regions of the IeDEA cohort (International epidemiology Databases to Evaluate AIDS).

DETAILED DESCRIPTION:
With the expansion of access to Anti-Retroviral Treatment (ART) in Low and Middle-Income Countries (LMIC), there is an increase in HIV drug resistance. The previously recommended 1st-line regimen of Tenofovir, Emtricitabine and Efavirenz (TEE) contains three drugs with a low genetic barrier to resistance. As a result, acquired drug resistance mutations are detected in the majority of people on TEE across different regions and HIV-1 subtypes. There has also been a steady increase in Pre-treatment Drug Resistance (PDR) as ART coverage has expanded in LMIC. WHO now recommends the use of Dolutegravir (DTG) in 1st -, 2nd and 3rd-line ART for adults and adolescents. Therefore, in most countries, PLHIV are transitioned to a DTG-based regimen. DTG is a potent Integrase Strand Transfer Inhibitor (InSTI) which has better efficacy and safety profile than Efavirenz in 1st-line therapy and Lopinavir/Ritonavir in 2nd-line therapy. DTG has a high genetic barrier to resistance, and resistance in ART-naïve individuals treated with combination ART has so far been rare. However, when used as monotherapy, or in people with pre-existing InSTI resistance, DTG is associated with a higher risk of virologic failure and resistance.

In this study, the investigators aim to -

1. Identify novel mutations or novel combinations of DTG Drug Resistance Mutations (DRMs).
2. Identify risk factors for virologic failure, development of InSTI DRMs and InSTI drug resistance.
3. Check the correlations between novel resistance genotypes and phenotypic DTG resistance across HIV-1 subtypes.

Adults (≥18 years) and adolescents (10-17 years) with virologic failure (viral load ≥1000 copies/mL) on any DTG-based anti-retroviral treatment (1st-line, 2nd-line and 3rd-line) at 20-30 clinical sites within six regions of the IeDEA cohort will be recruited into the study. There is only one study visit per participant and the study is observational and embedded in routine care, with no additional interventions. After obtaining informed consent, a blood specimen will be taken from the study participants. Whole genome sequencing will be performed using the Illumina MiSeq platform to identify the Drug Resistance Mutations. In addition, new DRMs and mutation pathways will be explored by viral genome-wide association study and conjunctive Bayesian network approaches.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older and adolescents (10-17 years)
* On any DTG-based ART regimen
* Who develop virologic failure (VF) defined as a VL >1000 copies/mL (single or confirmed measurement),
* and have signed the informed consent.

Exclusion Criteria:

* No Informed Consent

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients routinely treated at the local HIV care clinics.
Sampling Method: Probability Sample
Enrollment: 1103 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Type of Integrase Drug Resistance Mutations (INSTI DRMs) at the time of failing a DTG-based regimen. | 4 years
  The investigators define INSTI DRMs as all mutations associated with INSTIs by the Stanford HIVdb algorithm (https://hivdb.stanford.edu/). The identified mutations will be classified into major, accessory and other mutation types. New mutations will also be assessed. Analyses will be cross-sectional and differences between groups (for example, HIV-1 subtypes) tested using Pearson's chi-squared tests.
Prevalence of Integrase Drug Resistance Mutations (INSTI DRMs) at the time of failing a DTG-based regimen. | 4 years
  Prevalence of the identified mutations will be expressed as the proportion of the study population showing INSTI DRMs compared to the total number of study participants experiencing treatment failure (Viral load > 1000 copies/mL and successfully sequenced). Analyses will be cross-sectional and differences between groups (for example, HIV-1 subtypes) tested using Pearson's chi-squared tests.
Time to virologic failure | 4 years
  The Investigators define virologic failure as two consecutive viral load measurements of >1000 copies/mL of blood. The time to virologic failure will be analysed using survival models, stratified by country to account for heterogeneity, including all individuals who started Antiretroviral Therapy (ART) on a dolutegravir-based regimen or switched to such a regimen.
Number of INSTI DRMs per patient | 4 years
  The Investigators define INSTI DRMs as all mutations associated with INSTIs by the Stanford HIVdb algorithm, including major and accessory mutations (HIV Drug Resistance Database (https://hivdb.stanford.edu/)). All individuals who developed virologic failure on any dolutegravir-based regimen will be analysed using a negative binomial generalised linear model for the number of major/accessory INSTI DRMs per patient.
DTG drug resistance | 4 years
  The Investigators will use the Stanford HIV Database and the Stanford HIVdb algorithm (HIV Drug Resistance Database (https://hivdb.stanford.edu/)) to categorise drug resistance levels as susceptible (score below 10), potential low (10-14), low (15-29), intermediate (30-59), or high (≥60). An ordinal logistic regression model will be used to analyse the drug resistance levels.
Phenotypic resistance levels of novel DRMs | 1 year
  Selected samples will undergo phenotypic testing to identify any correlations between the observed DRMs on HIV phenotype, which is quantified as the fold change of IC50 to DTG, i.e. the concentration at which viral replication is reduced by 50%.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Egger, Prof. Dr., Study Director — Institute of Social and Preventive Medicine (ISPM), University of Bern, Switzerland; Richard Lessells, Dr., Principal Investigator — KwaZulu-Natal Research Innovation & Sequencing Platform, University of KwaZulu-Natal, South Africa; Roger Kouyos, Prof. Dr., Principal Investigator — Department of Infectious Diseases and Hospital Epidemiology, University of Zürich, Switzerland; Jonathan Sterne, Prof. Dr., Principal Investigator — University of Bristol; Niko Beerenwinkel, Prof. Dr., Principal Investigator — ETH Zurich (Switzerland)
Locations (22):
- Centro Medico Huesped, Buenos Aires, Argentina
- Instituto Nacional de Infectiologia Evandro Chagas - Fiocruz, Rio de Janeiro, Brazil
- Hopital de Jour du Centre Hospitalier Universitaire (CHU Souro Sanou), Bobo-Dioulasso, Burkina Faso
- National Centre for HIV/AIDS, Dermatology and STDs (NCHADS), Phnom Penh, Cambodia
- Cameroon (2):
  - Regional Hospital Limbe, Limbe
  - Hospital Jamot, Yaoundé
- Côte d’Ivoire (2):
  - ACONDA Centre de Prise en Charge et de Formation (CePReF), Abidjan
  - Centre médical de suivi des donneurs de sang, CNTS, Abidjan
- Moi University, AMPATH, Eldoret, Kenya
- Malawi (2):
  - Lighthouse clinic, Lilongwe
  - Martin Preuss Centre, Lilongwe
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico
- Republic of the Congo (2):
  - Centre de Traitement Ambulatoire, Brazzaville
  - Centre de Traitement Ambulatoire, Pointe-Noire
- Research for Development, Einstein-Rwanda Research and Capacity Building Program, Kigali, Rwanda
- National Institute for Medical Research (NIMR), Kisesa, Tanzania
- Thailand (2):
  - HIV-NAT/Thai Red Cross AIDS Research Center (TRCARC), Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
- Uganda (2):
  - Masaka Regional Referral Hospital / AHF Uganda Cares, Masaka
  - Mbarara University of Science and Technology / Mbarara ISS Clinic (MUST), Mbarara
- Centre for Infectious Disease Research Zambia (CIDRZ), Lusaka, Zambia
- Newlands Clinic, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
The Investigators are open to share any type of study data upon reasonable request, pending approval by local sites.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Within 1 year of study conclusion, for about 1 year.
Access Criteria: Upon reasonable request, pending approval by local sites.

REFERENCES:
- [Derived] Egger M, Sauermann M, Loosli T, Hossmann S, Riedo S, Beerenwinkel N, Jaquet A, Minga A, Ross J, Giandhari J, Kouyos RD, Lessells R. HIV-1 subtype-specific drug resistance on dolutegravir-based antiretroviral therapy: protocol for a multicentre study (DTG RESIST). BMJ Open. 2024 Aug 21;14(8):e085819. doi: 10.1136/bmjopen-2024-085819. PMID 39174068
- [Derived] Egger M, Sauermann M, Loosli T, Hossmann S, Riedo S, Beerenwinkel N, Jaquet A, Minga A, Ross JL, Giandhari J, Kouyos R, Lessells R. HIV-1 subtype-specific drug resistance on dolutegravir-based antiretroviral therapy: protocol for a multicentre longitudinal study (DTG RESIST). medRxiv [Preprint]. 2024 May 24:2024.05.23.24307850. doi: 10.1101/2024.05.23.24307850. PMID 38952780